CLINICAL TRIAL: NCT00328653
Title: Phase II/III, Multicenter, Double-Masked, Randomized, Parallel Group, Dose Ranging, Controlled Trial of Efficacy and Tolerance of Nova22007 (Cyclosporine A [CSA] 0.05% & 0.1% Ophthalmic Cationic Emulsion) Versus Vehicle in Patients With VKC
Brief Title: Efficacy and Tolerance of Nova22007 Versus Vehicle in Patients With Vernal Keratoconjunctivitis (VKC)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Santen SAS (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NOVATIVE - NVG05L101
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Conjunctivitis, Vernal
Keywords: vernal keratoconjunctivitis (VKC), eye, allergy, cyclosporin
MeSH Terms: conditions — Conjunctivitis, Allergic; Hypersensitivity

ARMS (3):
- NOVA22007 0.05% (Experimental): four times daily
  Interventions: Drug: Cyclosporine NOVA22007 0.05%
- NOVA22007 0.1% (Experimental): four times daily
  Interventions: Drug: Cyclosporine NOVA22007 0.1%
- Vehicle (Sham Comparator): administered four times daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Cyclosporine NOVA22007 0.05%
  Arms: NOVA22007 0.05%
Drug: Cyclosporine NOVA22007 0.1%
  Arms: NOVA22007 0.1%
Drug: Vehicle
  Arms: Vehicle

SUMMARY:
The primary objective of this study is:

* To assess the efficacy of Nova22007, a cyclosporine A (CsA), 0.05% and 0.1% versus vehicle in patients with vernal keratoconjunctivitis (VKC) after a 4-week treatment period.

The secondary objectives of this study are:

* To compare the safety and ocular tolerance of Nova22007 0.05% and 0.1%;
* To assess the long term safety and ocular tolerance of Nova22007 0.05% and 0.1%; and
* To assess the decrease in frequency of concomitant artificial tears use.

ELIGIBILITY:
Inclusion Criteria:

* At least the two following signs, in at least one eye* (the same eye should fulfill both criteria):

  * Presence of giant papillae with a diameter ≥ 1 mm on the upper tarsal conjunctiva AND
  * Superficial keratitis
* At least two of the following ocular symptoms with a score > 2 in at least one eye*: burning/stinging, tearing, itching, pain, sticky eyelids, foreign body sensation, mucus discharge, and photophobia.
* Hyperemia score equal to or greater than 2.

Exclusion Criteria:

* Concomitant corneal ulcer of infectious origin.
* Active ocular herpes
* Disease that could possibly interfere with the interpretation of the study results: active uveitis (defined by Tyndall score > 0), previous history of ocular hypertension or glaucoma, or condition incompatible with the frequent assessments needed by the study.
* Active herpes.
* History of malignancy or a recurrence in the last 5 years.
* Abnormality of nasolacrimal drainage apparatus.
* Concomitant disease not stabilized within 1 month before Screening Visit (e.g. diabetes with glycemia out of range, trouble with thyroid secretions, etc.) or judged by the investigator to be incompatible with the study (e.g. current systemic infections), or condition incompatible with the frequent assessments needed by the study.
* Known hypersensitivity to one of the components of the investigational medicinal products (IMP) or test products.
* Severe systemic allergy requiring systemic treatment at study entry.
* Female of childbearing potential.
* History of drug or alcohol addiction (> 50g/day, 5 glasses alcohol/day).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2006-05; Primary Completion 2007-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David BenEzra, Pf, Principal Investigator — Haddassah University Hospital; Christophe Baudouin, Pf., Study Director — Hôpital des XV-XX 28 rue de Charenton 75012 Paris
Locations (1):
- Groupe Hospitalier Bichat-Claude Bernard, Paris, France

REFERENCES:
- [Derived] Leonardi A, Pisella PJ, Benitez-Del-Castillo JM, Amrane M, Ismail D, Doan S, Bremond-Gignac D. NOVATIVE: A Phase II/III, Multicenter, Double-masked, Randomized Study of Cyclosporine A 0.05% and 0.1% Ophthalmic Cationic Emulsion Versus Vehicle in Patients with Vernal Keratoconjunctivitis. Clin Ther. 2023 Dec;45(12):1284-1288. doi: 10.1016/j.clinthera.2023.09.022. Epub 2023 Oct 21. PMID 37872059

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle: Vehicle administered four times daily
- NOVA22007 0.05%: Cyclosporine NOVA22007 0.05% four times daily
- NOVA22007 0.1%: Cyclosporine NOVA22007 0.1% four times daily
Period: Period I
Arm/Group | Vehicle | NOVA22007 0.05% | NOVA22007 0.1%
Started | 40 | 39 | 39
Completed | 36 | 39 | 36
Not Completed | 4 | 0 | 3
Period: Period II
Arm/Group | Vehicle | NOVA22007 0.05% | NOVA22007 0.1%
Started | 0 (Following completion of the first period of the trial, all patients were to be administered NOVA22007 (i.e. CsA 0.05% or 0.1%) as four times or twice daily instillations in both eyes for an additional 3 month period.) | 58 | 53
Completed | 0 | 50 | 49
Not Completed | 0 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NOVA22007 0.05% | NOVA22007 0.1% | Vehicle | Total
Number analyzed (Participants) | 39 | 39 | 40 | 118
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 8.5 (2.9) | 9.4 (3.7) | 8.5 (2.4) | 8.8 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11 | 22
  Male | 34 | 33 | 29 | 96

OUTCOME MEASURES:

1. Primary Outcome: Overall Rating of Subjective Symptoms of VKC in Period I
Description: The primary criteria of the trial was the overall rating of subjective symptoms in ocular symptoms of VKC as compared to Baseline and assessed at Week 4 (Month 1) based on a five-point scale based on BenEzra trial (BenEzra 1986):
  1. = Overall worsening of the subjective findings.
  2. = No change in the symptoms.
  3. = Slight improvement with the child still unable to participate in all normal daily activities.
  4. = Marked improvement despite temporary mild itching or mucus discharge.
  5. = Completely free of all symptoms.
Time Frame: Week 4
Population: FAS population
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | NOVA22007 0.05% | NOVA22007 0.1%
Number analyzed (Participants) | 40 | 39 | 39
Participants
  1- Overall worsening of the | 7 | 1 | 4
  2- No change in the symptoms | 5 | 3 | 2
  3- Slight improvement | 10 | 15 | 11
  4- Marked improvement | 15 | 19 | 20
  5- Completely free of all symptoms | 3 | 1 | 2
Statistical Analysis 1: Comparison: Vehicle vs NOVA22007 0.05%; Test type: Superiority — Comparisons of NOVA22007 0.05% to vehicle; p = 0.2699, Cochran-Mantel-Haenszel; M-H Chi-square = 1.2187
Statistical Analysis 2: Comparison: Vehicle vs NOVA22007 0.1%; Test type: Superiority — Comparisons of NOVA22007 0.1% to vehicle; p = 0.2719, Cochran-Mantel-Haenszel; M-H Chi-square = 1.2359

2. Secondary Outcome: Change in Mean Daily Number of Unpreserved Artificial Tears Instillations in Period I
Time Frame: Up to Month1
Population: The number of participants is reduced due to missing data.
Measure: Mean (Standard Deviation); unit: instillations
Arm/Group | Vehicle | NOVA22007 0.05% | NOVA22007 0.1%
Number analyzed (Participants) | 40 | 39 | 39
instillations
  Week1- Baseline: number analyzed (Participants) | 21 | 23 | 18
  Week1- Baseline | -0.5 (1.5) | 0.1 (2.2) | -0.1 (1.3)
  Week2- Baseline: number analyzed (Participants) | 20 | 27 | 17
  Week2- Baseline | -0.2 (0.9) | -0.4 (1.4) | -0.2 (1.5)
  Month1-Baseline: number analyzed (Participants) | 20 | 27 | 18
  Month1-Baseline | -0.4 (1.9) | -0.5 (1.5) | 0.0 (1.9)

3. Secondary Outcome: Ocular Tolerance in Period I
Description: Are the tested eye drops (other than concomitant tear substitute ) comfortable?
Time Frame: Up to Month1
Population: The number of participants is reduced due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | NOVA22007 0.05% | NOVA22007 0.1%
Number analyzed (Participants) | 40 | 39 | 39
Participants
  Week1: number analyzed (Participants) | 38 | 35 | 38
  Week1: No | 3 | 11 | 4
  Week1: Yes | 35 | 24 | 34
  Week2: number analyzed (Participants) | 37 | 38 | 37
  Week2: No | 3 | 5 | 6
  Week2: Yes | 34 | 33 | 31
  Month1: number analyzed (Participants) | 36 | 39 | 36
  Month1: No | 2 | 8 | 7
  Month1: Yes | 34 | 31 | 29

4. Primary Outcome: Overall Rating of Objective Symptoms of VKC in Period I
Description: Overall rating of objective signs was to be assessed under the slit lamp by the Investigator and recorded on a five-point scale based on BenEzra trial (BenEzra 1986):
  1. Intense congestion of conjunctival vessels, perilimbal injection, or corneal involvement with the papillary proliferations more extensive or similar to the situation recorded before treatment in at least one of the eyes.
  2. The overall condition was assessed as better than before treatment in both eyes.
  3. Total re-epithelialisation of the cornea although slight conjunctival and perilimbal hyperaemia and papillary proliferations remains in both eyes.
  4. Only slight conjunctival hyperaemia without perilimbal injection or papillary proliferations in at least one eye
  5. Both eyes were quiet with no papillary proliferations or conjunctival or perilimbal injection.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | NOVA22007 0.05% | NOVA22007 0.1%
Number analyzed (Participants) | 40 | 39 | 39
Participants
  1.Intense congestion of conjunctival vessels, perilimbal injection, or corneal involvement. | 18 | 8 | 7
  2.The overall condition was assessed as better than before treatment in both eyes. | 13 | 17 | 16
  3.Total re-epithelialisation of the cornea | 4 | 7 | 12
  4.Only slight conjunctival hyperaemia in at least one eye | 4 | 6 | 2
  4.Both eyes were quiet with no papillary proliferations or conjunctival or perilimbal injection. | 1 | 1 | 2
Statistical Analysis 1: Comparison: Vehicle vs NOVA22007 0.05%; Test type: Superiority — Comparisons of NOVA22007 0.05% to vehicle; p = 0.0386, Cochran-Mantel-Haenszel; M-H-Chi-square = 4.2925
Statistical Analysis 2: Comparison: Vehicle vs NOVA22007 0.1%; Test type: Superiority — Comparisons of NOVA22007 0.1% to vehicle; p = 0.0208, Cochran-Mantel-Haenszel; M-H-Chi-square = 5.3007

ADVERSE EVENTS:
Time Frame: From the time the patient gave informed consent until the last trial visit at month 4.
Groups:
- Period I- NOVA22007 0.05%: Low Dose Regimen
- Period I-NOVA22007 0.1%: High Dose Regimen
Arm/Group | Placebo | Period I- NOVA22007 0.05% | Period I-NOVA22007 0.1% | Period II- NOVA22007 0.05% | Period II-NOVA22007 0.1%
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39 | 0/39 | 0/58 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39 | 0/39 | 1/58 | 0/53
Other Adverse Events (participants affected / at risk) | 14/40 | 14/39 | 12/39 | 17/58 | 11/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | Period I- NOVA22007 0.05% (N=39) | Period I-NOVA22007 0.1% (N=39) | Period II- NOVA22007 0.05% (N=58) | Period II-NOVA22007 0.1% (N=53)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | Period I- NOVA22007 0.05% (N=39) | Period I-NOVA22007 0.1% (N=39) | Period II- NOVA22007 0.05% (N=58) | Period II-NOVA22007 0.1% (N=53)
Allergic keratitis (Eye disorders) | 9 | 3 | 8 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 3 | 3 | 1
Ocular hyperaemia (Eye disorders) | 1 | 2 | 2 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Corneal Epithelium disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0
Corneal neovascularisation (Eye disorders) | 0 | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 1 | 0
Instillation site pain (General disorders) | 2 | 0 | 1 | 0 | 1
Instillation site pruritus (General disorders) | 1 | 5 | 4 | 3 | 1
Drug intolerance (General disorders) | 0 | 2 | 0 | 4 | 1
Hyperthermia (General disorders) | 0 | 1 | 0 | 0 | 0
Instillation site lacrimation (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Corneal Ulcer (Eye disorders) | 3 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Instillation Site Irritation (General disorders) | 0 | 4 | 2 | 2 | 4
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes